CLINICAL TRIAL: NCT04510025
Title: Assessing the Effects of Coronavirus Disease (COVID-19) on Multiple Organ Systems and Impact on Quality of Life, Functional Capacity and Mental Health
Brief Title: Capturing MultiORgan Effects of COVID-19
Acronym: C-MORE
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 282608
Record Dates: First submitted 2020-07-14; First posted 2020-08-12 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Coronavirus Infection; Multi-Organ Disorder
Keywords: Coronavirus disease; MRI; Multi-organ injury; Quality of Life; Mental Health
MeSH Terms: conditions — Coronavirus Infections; Psychological Well-Being | interventions — Magnetic Resonance Imaging; Exercise Test; Spirometry; Walk Test; Hematologic Tests; Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 ml of blood stored
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-COVID: We will enrol age, gender, BMI and co-morbidity matched non-COVID control subjects (no serological evidence of previous infection, or active/previous symptoms suggestive of COVID-19). A minimum of 200 controls (as part of the COSMIC study) will be recruited.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- COVID-19: Hospitalised patients with moderate to severe infection (admitted for at least 2 days in hospital).
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — We will undertake multi-organ MRI to assess the health of vital organs including the brain, heart, lung, kidneys and liver. We will additionally examine the burden of ongoing respiratory limitations, mental health problems and quality of life in survivors of COVID-19 at 3, 6 and 12 months.
  Other Names: Cardiopulmonary exercise test; Spirometry; 6 minute walk test; Questionnaires (mental health, cognitive assessment and quality of life); Blood test; Transthoracic echocardiography (Sub-study); CT lungs (Sub-study)

SUMMARY:
The C-MORE study is prospective observational holistic longitudinal study which will characterise the prevalence of multi-organ injury among COVID-19 survivors post hospital discharge and assess its effects on quality of life, exercise tolerance and mental health.

DETAILED DESCRIPTION:
Since the outbreak of Coronavirus disease (COVID-19), hundreds of thousands of lives have been lost and millions significantly affected. Although primarily a respiratory viral illness, emerging data suggests that multiorgan involvement is common in those with moderate-severe infections. Whether or not persistent multiorgan damage will be seen in COVID-19 survivors is unknown.

C-MORE is an observational study that aims to investigate the long-term effects of COVID-19 on the lungs, heart, brain, liver and kidneys using advanced state-of-the art magnetic resonance imaging (MRI) technology. The study will assess 616 patients with laboratory-confirmed COVID-19 from leading UK centres and undertake multi-organ magnetic resonance imaging at 3, 6, and 12 months following the onset of COVID-19 symptoms. In addition, assessments of breathing, exercise capacity, cognition and mental health will be carried out.

The study will describe the prevalence of persistent multi-organ injury in COVID-19 patients and assess how this relates to comorbid conditions, severity of acute respiratory illness, immunological response, genetic factors, quality of life and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosis of COVID-19 infection confirmed by detection of viral nucleic acid on reverse-transcription Polymerase Chain Reaction (RT-PCR).
* Infection should be of moderate to severe intensity (i.e, patients with clinical signs of pneumonia such as respiratory rate > 30 breaths/min; or severe respiratory distress; or SpO2 < 90% (on room air) and admission for >48 hours.
* Controls: Participants with no serological evidence of previous infection, or active/previous symptoms suggestive of COVID-19, and who may or may not have comorbidities.

Exclusion Criteria:

* Contraindication to MRI e.g. pregnancy, pacemaker, ferromagnetic implant, shrapnel injury, severe claustrophobia, inability to lie flat.
* Any other significant disease or disorder which, in the opinion of the investigator, might influence the participant's ability to participate in the study.
* Any signs of active COVID-19 infection on day of visit.
* Significantly impaired renal function (eGFR<30 ml/min)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 500 participants who have recently been hospitalised with moderate-severe COVID-19 infection.
  A minimum of 200 individuals with no serological evidence of previous infection , or active/previous symptoms suggestive of COVID-19 will serve as controls.
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2020-05-13 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of damage (quantitative measures of injury) on lung, heart, liver, kidneys and brain MRI. | 6 months
  Characterise and compare the prevalence and extent of lung, heart, liver, kidney, brain injury on magnetic resonance imaging (MRI) in patients with moderate to severe COVID-19 disease with matched uninfected controls.

SECONDARY OUTCOMES:
Prevalence of damage (quantitative measures of injury) on lungs, heart, liver, kidneys and brain on MRI. | 3 and 12 months
  Characterise and compare the prevalence and extent of lung, heart, liver and kidney, brain injury on magnetic resonance imaging (MRI) in patients with moderate to severe COVID-19 disease with matched uninfected controls.
Prevalence of acute/chronic cardiac, renal and liver injury on blood tests. | 3, 6,12 months
  Characterise and compare the prevalence of cardiac, renal and liver injury on blood test in COVID-19 survivors and controls.
VO2 max on cardiopulmonary exercise testing | 3, 6,12 months
  Characterise and compare VO2 max on cardiopulmonary exercise testing in COVID-19 survivors and controls.
Prevalence of abnormal lung function test (any of the following: Forced expiratory volume in 1 second (FEV1)< 80% of predicted FEV1, or forced vital capacity (FVC)<80% predicted, ratio of FEV1/FVC >0.7 or diffusion lung capacity (<80% predicted)) | 3, 6,12 months
  Characterise and compare the prevalence of lung function test abnormalities among survivors and controls.
Quality of life - Short form-36 SF-36 score | 3, 6,12 months
  For each of the eight domains that the SF36 measures an aggregate percentage score is produced. The percentage scores range from 0% (lowest or worst possible level of functioning) to 100% (highest or best possible level of functioning).
Prevalence of impaired cognitive function on Montreal Cognitive assessment (MoCA<26) | 3, 6,12 months
  Described and compare the prevalence of impaired cognition (MoCA) between COVID-19 survivors and controls. MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
6-minute walk distance | 3, 6,12 months
  Compare 6-minute walk distance between COVID-19 survivors and controls.
Severity of anxiety on GAD-7 (Score) | 3, 6,12 months
  Compare prevalence and severity of anxiety between COVID-19 survivors and controls.
Severity of depression on PHQ-9 (Score) | 3, 6,12 months
  Compare prevalence and severity of depression among COVID-19 survivors and controls. PHQ-9 total score for the nine items ranges from 0 to 27. Scores of 5, 10, 15, and 20 represent outpoints for mild, moderate, moderately severe and severe depression, respectively.
Association between the extent of multi-organ injury (continuous variable) and markers of inflammation (white cell count). | 3,6,12 months
  To assess the association of multi organ damage on MRI and inflammatory response.
Correlation between the extent of symptoms (dyspnoea-12 score and fatigue score) and multi-organ injury. | 3,6,12months.
  To assess the association of ongoing symptomatology and multi-organ injury/inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shergill S, Elshibly M, Hothi SS, Parke KS, England RJ, Wormleighton JV, Hudson GJ, Tunnicliffe EM, Wild J, Smith SM, Francis S, Toshner M, Sattar N, Khunti K, Brightling CE, Antoniades C, Berry C, Greenwood JP, Moss A, Neubauer S, McCann GP, Raman B, Arnold JR. Assessing the impact of COmorbidities and Sociodemographic factors on Multiorgan Injury following COVID-19: rationale and protocol design of COSMIC, a UK multicentre observational study of COVID-negative controls. BMJ Open. 2025 Mar 6;15(3):e089508. doi: 10.1136/bmjopen-2024-089508. PMID 40050066
- [Derived] C-MORE/PHOSP-COVID Collaborative Group. Multiorgan MRI findings after hospitalisation with COVID-19 in the UK (C-MORE): a prospective, multicentre, observational cohort study. Lancet Respir Med. 2023 Nov;11(11):1003-1019. doi: 10.1016/S2213-2600(23)00262-X. Epub 2023 Sep 22. PMID 37748493
- See also: Interim results — https://pmc.ncbi.nlm.nih.gov/articles/PMC7615263/